CLINICAL TRIAL: NCT04975308
Title: EMBER-3: A Phase 3, Randomized, Open-Label Study of Imlunestrant, Investigator's Choice of Endocrine Therapy, and Imlunestrant Plus Abemaciclib in Patients With Estrogen Receptor Positive, HER2 Negative Locally Advanced or Metastatic Breast Cancer Previously Treated With Endocrine Therapy
Brief Title: A Study of Imlunestrant, Investigator's Choice of Endocrine Therapy, and Imlunestrant Plus Abemaciclib in Participants With ER+, HER2- Advanced Breast Cancer
Acronym: EMBER-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18175; J2J-OX-JZLC (Other: Eli Lilly and Company); 2021-000079-35 (EudraCT Number); 2023-506786-63-00 (EU CTIS Number)
Record Dates: First submitted 2021-07-22; First posted 2021-07-23 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: SERD
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Imlunestrant; exemestane; Fulvestrant; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Imlunestrant (Experimental): Participants received Imlunestrant 400 milligrams (mg) orally once daily on days 1 to 28 of a 28-day cycle, until disease progression or a criterion for discontinuation were met.
  Interventions: Drug: Imlunestrant
- Arm B: Investigator's Choice of Endocrine Therapy (Experimental): Participants received the investigator's choice of endocrine therapy, either exemestane 25 mg administered orally once daily on days 1 to 28 of a 28-day cycle, or Fulvestrant 500 mg intramuscularly on days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond, until disease progression or a criterion for discontinuation was met.
  Interventions: Drug: Exemestane; Drug: Fulvestrant
- Arm C: Imlunestrant + Abemaciclib (Experimental): Participants received Imlunestrant 400 mg orally once daily on Days 1 to 28 of a 28-day cycle, plus Abemaciclib 150 mg orally twice daily on Days 1 to 28 of a 28-day cycle, until disease progression or a criterion for discontinuation was met.
  Interventions: Drug: Imlunestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Imlunestrant — Administered orally.
  Other Names: LY3484356
  Arms: Arm A: Imlunestrant; Arm C: Imlunestrant + Abemaciclib
Drug: Exemestane — Administered orally.
  Arms: Arm B: Investigator's Choice of Endocrine Therapy
Drug: Fulvestrant — Administered IM.
  Arms: Arm B: Investigator's Choice of Endocrine Therapy
Drug: Abemaciclib — Administered orally.
  Other Names: LY2835219
  Arms: Arm C: Imlunestrant + Abemaciclib

SUMMARY:
The main purpose of this study is to measure how well imlunestrant works compared to standard hormone therapy, and how well imlunestrant with abemaciclib work compared to imlunestrant in participants with breast cancer that is estrogen receptor positive (ER+) and human epidermal receptor 2 negative (HER2-). Participants must have breast cancer that is advanced or has spread to another part of the body. Study participation could last up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of ER+, HER2- locally advanced or metastatic breast cancer
* Have disease that has demonstrated progression on or after an aromatase inhibitor alone or in combination with a cyclin-dependent kinase (CDK)4/6 inhibitor

  -- Participants are expected to have received prior treatment with a CDK4/6 inhibitor, if this treatment is approved and can be reimbursed
* Must be deemed appropriate for treatment with endocrine therapy
* If female, have a postmenopausal status by natural or surgical means or by ovarian function suppression
* Have RECIST evaluable disease (measurable disease and/or nonmeasurable bone-only disease)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group scale (Oken et al. 1982)
* Have adequate renal, hematologic, and hepatic organ function
* Must be able to swallow capsules/tablets

Exclusion Criteria:

* Have received prior treatment with chemotherapy (except for neoadjuvant/ adjuvant chemotherapy), fulvestrant, or any investigational-ER-directed therapy (including SERDs and non-SERDs), any PI3K-, mTOR- or AKT- inhibitor
* Have visceral crisis, lymphangitic spread within the lung, or any evidence of leptomeningeal disease.
* Have symptomatic or untreated brain metastasis.
* Have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study
* Known allergic reaction against any of the components of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 874 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2027-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (243):
- United States (48):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Marin Cancer Care, Greenbrae, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - Banner MD Anderson Cancer Center at McKee Medical Center, Loveland, Colorado
  - Clermont Oncology Center, Clermont, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem - Evanston Hospital, Evanston, Illinois
  - IU Health Ball Memorial Hospital, Inc., Muncie, Indiana
  - The University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Care Access - Clifton, Clifton, New Jersey
  - Memorial Sloan Kettering - Bergen, Montvale, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - Avera Cancer Institute Sioux Falls, Sioux Falls, South Dakota
  - Florida Cancer Specialists, Nashville, Tennessee
  - The Mark H Zangmeister Cancer Center, Nashville, Tennessee
  - USO - Texas Oncology - Allen, Allen, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Willamette Valley Cancer Institute & Research Ctr., Houston, Texas
  - Texas Oncology - Carrollton, Lewisville, Texas
  - Texas Oncology - Denison, The Woodlands, Texas
  - Texas Oncology - Paris, The Woodlands, Texas
  - Blue Ridge Cancer Care, The Woodlands, Texas
  - Broome Oncology, The Woodlands, Texas
  - Minnesota Oncology/Hematology PA, The Woodlands, Texas
  - Texas Oncology - Carrollton, The Woodlands, Texas
  - Texas Oncology - McKinney, The Woodlands, Texas
  - Texas Oncology - Medical City Dallas, The Woodlands, Texas
  - Texas Oncology - Methodist Charlton Cancer Center, The Woodlands, Texas
  - Texas Oncology - San Antonio Medical Center, The Woodlands, Texas
  - Texas Oncology - The Woodlands, The Woodlands, Texas
  - Texas Oncology - Willowbrook, The Woodlands, Texas
  - Texas Oncology Fort Worth, The Woodlands, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, The Woodlands, Texas
  - USO-Rocky Mountain Cancer Center, The Woodlands, Texas
  - Texas Oncology - Austin Central, The Woodlands, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - The University of Vermont Medical Center Inc., Burlington, Vermont
- Argentina (8):
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - CIPREC, Buenos Aires, Buenos Aires F.D.
  - Fundación Cenit Para La Investigación En Neurociencias, CABA, Buenos Aires F.D.
  - Centro Medico Privado CEMAIC, Capital, Córdoba Province
  - Clinica Viedma, Viedma, Río Negro Province
  - Instituto Argentino de Diagnóstico y Tratamiento (IADT), Buenos Aires
  - Instituto San Marcos, San Juan
  - Sanatorio Norte, Santiago del Estero
- Australia (5):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Maroondah Hospital, Melbourne, Victoria
- Austria (3):
  - Medizinische Universität Graz, Graz, Styria
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna, Vienna
  - Uniklinikum Salzburg, Salzburg
- Belgium (8):
  - Imelda General Hospital, Bonheiden, Antwerpen
  - Institut Jules Bordet, Brussels, Bruxelles-Capitale, Région de
  - UZ Brussel, Brussels, Bruxelles-Capitale, Région de
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Nikolaas, Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Groeninge Campus Kennedylaan, Kortrijk, West-Vlaanderen
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
- Brazil (5):
  - Hospital de Cancer de Londrina, Londrina, Paraná
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Clínica de Pesquisa e Centro de Estudos em Ginecologia Oncológica e Mamária LTDA, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo, São Paulo
- China (31):
  - Afflilated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Centre, Guangzhou, Guangdong
  - Jiangmen Center Hospital, Jiangmen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Zhongshan Peoples Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-Sen University, Zhuhai, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Hwa Mei Hospital University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - Ningbo Medical Center, Ningbo, Zhejiang
- Czechia (5):
  - Nemocnice Horovice, Hořovice, Beroun
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha 10
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Nemocnice Na Bulovce, Prague, Praha 8
  - Oblastni nemocnice Pribram, Příbram, Příbram
- France (9):
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg, Alsace
  - Polyclinique De Blois, La Chaussée-Saint-Victor, Centre-Val de Loire
  - CHU Besançon, Besançon, Doubs
  - Hôpital René Huguenin, Saint-Cloud, Hauts-de-Seine
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-Roussillon
  - Clinique Victor Hugo Le Mans, Le Mans, Pays de la Loire Region
  - Centre Hospitalier de la Côte Basque, Bayonne, Pyrénées-Atlantiques
  - Institut Curie, Paris
  - Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (9):
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Onkologiezentrum Donauwörth, Donauwörth, Bavaria
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München, Bavaria
  - Agaplesion Markus Krankenhaus, Frankfurt am Main, Hesse
  - Gynäkologisch-Onkologische Praxis am Pelikanplatz, Hanover, Lower Saxony
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung, Essen, North Rhine-Westphalia
  - Evangelisches Krankenhaus Bethesda Mönchengladbach, Mönchengladbach, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
- Greece (8):
  - Agios Savvas Regional Cancer Hospital, Athens, Attikí
  - Alexandra Hospital, Athens, Attikí
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", Nea Kifissia, Attikí
  - University General Hospital of Heraklion, Heraklion, Irakleío
  - Euromedica General Clinic of Thessaloniki, Thessaloniki, Thessaloníki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki, Thessaloníki
  - European Interbalkan Medical Center, Thessaloniki, Thessaloníki
  - University General Hospital of Larissa, Larissa, Thessalía
- India (9):
  - Medstar Speciality Hospital, Bangalore, Karnataka
  - Regional Cancer Centre - Thiruvananthapuram, Thiruvananthapuram, Kerala
  - HCG Cancer Centre, Mumbai, Maharashtra
  - Government Medical College And Hospital - Nagpur, Nagpur, Maharashtra
  - Rashtrasant Tukdoji Regional Cancer Hospital, Nagpur, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Lifepoint Multispeciality Hospital, Pune, Maharashtra
  - Yashoda Hospitals, Hyderabad, Telangana
- Italy (7):
  - University of Naples Federico II, Naples, Campania
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli, Campania
  - Cro-Irccs, Aviano, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Ospedale San Martino, Genoa, Liguria
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Istituto Oncologico Veneto IRCCS, Padua
- Japan (22):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba cancer center, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume General Hospital, Kurume, Fukuoka
  - Gunma Prefectural Cancer Center, Otashi, Gunma
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Shinko Hospital, Kobe, Hyōgo
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaraki
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Nagano Municipal Hospital, Tomitake, Nagano
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Showa University Hospital, Shinagawa, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hospital, Hiroshima
  - Sagara Hospital, Kagoshima
  - Kumamoto Shinto General Hospital, Kumamoto
  - Osaka International Cancer Institute, Osaka
  - Shizuoka General Hospital, Shizuoka
  - Juntendo University Hospital, Tokyo
- Mexico (9):
  - Centro de Investigación Clínica de Alta Especialidad, Torreón, Coahuila
  - COI Centro Oncologico Internacional S.A.P.I. de C.V., Álvaro Obregón, Mexico City
  - Grupo Medico Camino Sc, Mexico City, Mexico City
  - Private Practice - Dr. Joaquin Reinoso, Monterrey, Nuevo León
  - Filios Alta Medicina, Monterrey, Nuevo León
  - Centro Medico Zambrano Hellion, San Pedro Garza García, Nuevo León
  - Unidad de Investigación en Salud, Chihuahua City
  - Oaxaca Site Management Organization, Oaxaca City
  - Unidad Médica Onco-hematológica, Puebla City
- Netherlands (3):
  - Maastricht UMC+, Maastricht, Limburg
  - Medische Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Haga Ziekenhuis locatie Leyweg, The Hague, South Holland
- Russia (3):
  - Kaluga Regional Clinical Oncology Center, Kaluga, Kalužskaja Oblast'
  - Volgograd Regional Clinical Cancer Clinic No.1, Volgograd, Volgograd Oblast
  - N.N.Petrov Research Institute of Oncology, Saint Petersburg
- South Korea (12):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan-si, Chungcheongnam-do [Chungnam]
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [Incheon]
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Yeungnam Univeristy Medical Center, Daegu, Kyǒngsangbuk-do
  - Dong-A University Hospital, Busan, Pusan-Kwangyǒkshi
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kangbuk Samsung Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Gangnam Severance Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kyungpook National University Chilgok Hospital, Daegu, Taegu-Kwangyǒkshi
- Spain (13):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitari Dexeusa, Barcelona, Catalunya [Cataluña]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [Cataluña]
  - Hospital San Pedro de Alcántara, Cáceres, Extremadura
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida, Lleida [Lérida]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Quirónsalud Valencia, Valencia, València
  - Hospital Universitario San Cecilio, Granada
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
- Taiwan (5):
  - Chi Mei Hospital - Liouying Branch, Tainan, Tainan
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
- Turkey (Türkiye) (16):
  - Medipol University Medical Faculty, Stanbul, Istanbul
  - Acibadem Altunizade Hospital, Üsküdar / Stanbul, Istanbul
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - University of Health Sciences,Gulhane School of Medicine, Ankara
  - Abdurrahman Yurtaslan Ankara Oncology, education and Research Hospital, Ankara
  - Hacettepe Universitesi, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Dicle Üniversitesi, Diyarbakır
  - Trakya University, Edirne
  - Acıbadem Maslak Hastanesi, Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Ege Universitesi Hastanesi, Izmir
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi, Malatya
  - Mersin University, Mersin
- Ukraine (5):
  - Communal Enterprise 'Kryvyi Rih Oncology Dispensary' of the Dnipropetrovsk Regional Council, Kryvyi Rih, Dnipropetrovsk Oblast
  - CNPE "Regional Center of Oncology", Kharkiv, Kharkivs’ka Oblast’
  - Municipal non-profit enterprise'Odesa Regional Clinical Hospital'of Odesa Regional Council, Odesa, Odesa Oblast
  - Municipal Enterprise "Volyn Regional Medical Oncology Centre" of the Volyn Regional Council, Lutsk, Volyn Oblast
  - Uzhgorod Central City Clinical Hospital, Uzhhorod, Zakarpattia Oblast

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Jhaveri KL, Neven P, Casalnuovo ML, Kim SB, Tokunaga E, Aftimos P, Saura C, O'Shaughnessy J, Harbeck N, Carey LA, Curigliano G, Llombart-Cussac A, Lim E, Garcia Tinoco ML, Sohn J, Mattar A, Zhang Q, Huang CS, Hung CC, Martinez Rodriguez JL, Ruiz Borrego M, Nakamura R, Pradhan KR, Cramer von Laue C, Barrett E, Cao S, Wang XA, Smyth LM, Bidard FC; EMBER-3 Study Group. Imlunestrant with or without Abemaciclib in Advanced Breast Cancer. N Engl J Med. 2025 Mar 27;392(12):1189-1202. doi: 10.1056/NEJMoa2410858. Epub 2024 Dec 11. PMID 39660834
- See also: Study of LY3484356 Versus Hormone Therapy, in Participants With Estrogen Receptor Positive (ER+), Human Epidermal Growth Factor Receptor 2 Negative (HER2-) Breast Cancer (EMBER-3) — https://trials.lilly.com/en-US/trial/297163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initially planned with participants randomized 1:1 to either arm A or arm B. Following a protocol amendment, arm C was added later, after randomization to arms A and B had already begun.
Period: Overall Study
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy | Arm C: Imlunestrant + Abemaciclib
Started | 331 | 330 | 213
Analysis Population for the Comparison Between Arm A and Arm B (All participants who were randomly assigned to either Arm A or Arm B.) | 331 | 330 (For analyses between Arm A and Arm B, the study was planned to analyze Arm B as a whole, regardless of whether the participants received exemestane or fulvestrant as the Investigator's Choice of Endocrine Therapy.) | 0
Analysis Population for the Comparison Between Arm C and Arm A (For analyses between arm C and arm A, the study was planned to include participants who were randomized to these arms concurrently.) | 213 | 0 | 213
Estrogen Receptor 1 (ESR1) Mutation-Detected Population for Comparison Between Arm A and Arm B | 138 | 118 | 0
Received at Least 1 Dose of Study Drug | 326 | 324 | 209
Safety Analysis Population (All randomised participants who received at least 1 dose of study drug. Participants were analyzed according to the study treatment they actually received.) | 327 (One participant assigned to Arm C received Imlunestrant alone (i.e., did not receive abemaciclib) and was therefore included in Arm A for safety analyses.) | 324 (Investigator's Choice of Endocrine Therapy: * exemestane = 32 * fulvestrant = 292) | 208
Completed (Participants with progressive disease or death were considered study completers.) | 246 | 264 | 117
Not Completed | 85 | 66 | 96
Not completed — Withdrawal by Subject | 6 | 16 | 6
Not completed — Physician Decision | 0 | 3 | 1
Not completed — Adverse Event | 10 | 1 | 12
Not completed — On study treatment (Ongoing) | 65 | 43 | 75
Not completed — Protocol Deviation | 4 | 3 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Imlunestrant: Participants received Imlunestrant 400 milligrams (mg) orally once daily on days 1 to 28 of a 28-day cycle, until disease progression or a criterion for discontinuation were met.
- Investigator's Choice of Endocrine Therapy: Participants received the investigator's choice of endocrine therapy, either exemestane 25 mg administered orally once daily on days 1 to 28 of a 28-day cycle, or Fulvestrant 500 mg intramuscularly on days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond, until disease progression or a criterion for discontinuation was met.
- Imlunestrant + Abemaciclib: Participants received Imlunestrant 400 mg orally once daily on Days 1 to 28 of a 28-day cycle, plus Abemaciclib 150 mg orally twice daily on Days 1 to 28 of a 28-day cycle, until disease progression or a criterion for discontinuation was met.
- Total: Total of all reporting groups
Arm/Group | Imlunestrant | Investigator's Choice of Endocrine Therapy | Imlunestrant + Abemaciclib | Total
Number analyzed (Participants) | 331 | 330 | 213 | 874
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.6) | 60.8 (12.0) | 61.9 (11.1) | 60.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 327 | 329 | 211 | 867
  Male | 4 | 1 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 80 | 37 | 196
  Not Hispanic or Latino | 218 | 216 | 148 | 582
  Unknown or Not Reported | 34 | 34 | 28 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 23 | 16 | 3 | 42
  Asian | 92 | 96 | 72 | 260
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 7 | 8 | 26
  White | 186 | 191 | 111 | 488
  More than one race | 2 | 7 | 3 | 12
  Unknown or Not Reported | 17 | 13 | 16 | 46
Estrogen Receptor 1 (ESR1)-Mutation [Count of Participants; unit: Participants]
  Detected | 138 | 118 | 67 | 323
  Not detected | 193 | 212 | 146 | 551

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Progression Free Survival (PFS) (Between Arm A and Arm B)
Description: PFS was defined as the time from randomization to the date of first documented progression of disease or death from any cause in the absence of disease progression using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria, as assessed by investigator. Progressive disease (PD) was defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Participants known to be alive and without disease progression were censored at the date of their last adequate tumor assessment per RECIST 1.1 criteria, or date of randomization (whichever is later).
Time Frame: Randomization to the date of first documented progression of disease or death from any cause (up to 28 months)
Population: All participants who were randomly assigned to either arm A or arm B (including censored). Number of participants censored in "Arm A=94," "Arm B=77."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 331 | 330
Months | 5.55 [5.32 to 7.26] | 5.52 [4.60 to 5.62]
Statistical Analysis 1: Comparison: Arm A: Imlunestrant vs Arm B: Investigator's Choice of Endocrine Therapy; Test type: Superiority; p = 0.1158, Log Rank; Hazard Ratio (HR) = 0.867, 95% CI 2-sided [0.724 to 1.039]

2. Primary Outcome: Investigator-assessed PFS (Between Arm C and Arm A)
Description: as for outcome 1
Time Frame: Randomization to the date of first documented progression of disease or death from any cause (up to 26 months)
Population: All participants who were randomly assigned to either arm A or arm C concurrently (including censored). Number of participants censored in "Arm C=99," "Arm A=64."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Imlunestrant + Abemaciclib | Arm A: Imlunestrant
Number analyzed (Participants) | 213 | 213
Months | 9.36 [7.49 to 11.86] | 5.49 [3.78 to 5.62]
Statistical Analysis 1: Comparison: Arm C: Imlunestrant + Abemaciclib vs Arm A: Imlunestrant; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.569, 95% CI 2-sided [0.441 to 0.733]

3. Primary Outcome: Investigator-assessed PFS in the Estrogen Receptor 1 (ESR1)-Mutation Detected Population (Between Arm A and Arm B)
Description: as for outcome 1
Time Frame: Randomization to the date of first documented progression of disease or death from any cause (up to 28 months)
Population: All participants who were randomly assigned to either arm A or arm B and had ESR1 mutations detected at baseline (including censored). Number of participants censored in "Arm A=29," "Arm B=16."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 138 | 118
Months | 5.49 [3.91 to 7.39] | 3.84 [3.68 to 5.52]
Statistical Analysis 1: Comparison: Arm A: Imlunestrant vs Arm B: Investigator's Choice of Endocrine Therapy; Test type: Superiority; p = 0.0008, Log Rank; Hazard Ratio (HR) = 0.617, 95% CI 2-sided [0.464 to 0.821]

4. Secondary Outcome: Blinded Independent Review Committee (BIRC) Assessed PFS (Between Arm A and Arm B)
Description: as for outcome 1
Time Frame: Randomization to the date of first documented progression of disease or death from any cause (up to 28 months)
Population: All participants who were randomly assigned to either arm A or arm B (including censored). Number of participants censored in "Arm A=171," "Arm B=171."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 331 | 330
Months | 9.23 [7.33 to 11.07] | 7.36 [5.55 to 9.40]

5. Secondary Outcome: Blinded Independent Review Committee (BIRC) Assessed PFS (Between Arm C and Arm A)
Description: as for outcome 1
Time Frame: Randomization to the date of first documented progression of disease or death from any cause (up to 25 months)
Population: All participants who were randomly assigned to either arm A or arm C concurrently (including censored). Number of participants censored in "Arm C=132," "Arm A=116."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Imlunestrant + Abemaciclib | Arm A: Imlunestrant
Number analyzed (Participants) | 213 | 213
Months | 14.52 [11.37 to NA] — Due to the high number of censored participants, there were not enough events to estimate the upper limit of the 95% confidence interval. | 9.23 [5.49 to 13.70]

6. Secondary Outcome: Percentage of Participants With Investigator-assessed Objective Response Rate (ORR) (Between Arm A and Arm B)
Description: ORR was the best confirmed overall tumor response of complete response (CR) or partial response (PR) as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions.
Time Frame: Randomization until measured progressive disease (up to 28 months)
Population: All participants who were randomly assigned to either arm A or arm B.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 331 | 330
Percentage of participants | 10.3 [7 to 13.5] | 6.4 [3.7 to 9]

7. Secondary Outcome: Investigator-assessed Duration of Response (DoR) (Between Arm A and Arm B)
Description: DoR is defined as the time from the date measurement criteria for CR or PR (whichever is first recorded) are first met until the first date that disease is recurrent or objective progression is observed, per RECIST 1.1 criteria, or the date of death from any cause in the absence of objectively determined disease progression or recurrence. Participants known to be alive and without disease progression were censored at the date of their last adequate tumor assessment per RECIST 1.1 criteria, or date of randomization (whichever is later).
Time Frame: From Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up To 26 Months)
Population: All participants who were randomly assigned to either arm A or arm B and had achieved CR or PR responses (including censored). Number of participants censored in "Arm A=17," "Arm B=7."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 34 | 21
Months | 11.10 [7.43 to 23.92] | 7.39 [5.59 to 15.67]

8. Secondary Outcome: Percentage of Participants With Investigator-assessed Clinical Benefit Rate (CBR) (Between Arm A and Arm B)
Description: CBR was the best confirmed overall tumor response of stable disease (SD) for greater than or equal to (≥) 24 weeks, CR or PR as defined by RECIST v1.1. CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Randomization until measured progressive disease (up to 28 months)
Population: All participants who were randomly assigned to either arm A or arm B.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 331 | 330
Percentage of participants | 46.8 [41.5 to 52.2] | 45.5 [40.1 to 50.8]

9. Secondary Outcome: Percentage of Participants With Investigator-assessed Objective Response Rate (ORR) (Between Arm C and Arm A)
Description: as for outcome 6
Time Frame: Randomization until measured progressive disease (up to 26 months)
Population: All participants who were randomly assigned to either arm A or arm C concurrently.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm C: Imlunestrant + Abemaciclib | Arm A: Imlunestrant
Number analyzed (Participants) | 213 | 213
Percentage of participants | 21.1 [15.6 to 26.6] | 9.4 [5.5 to 13.3]

10. Secondary Outcome: Investigator-assessed Duration of Response (DoR) (Between Arm C and Arm A)
Description: as for outcome 7
Time Frame: From Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up To 19 Months)
Population: All participants who were randomly assigned to either arm C or arm A and had achieved CR or PR responses (including censored). Number of participants censored in "Arm C=30," "Arm A=11."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Imlunestrant + Abemaciclib | Arm A: Imlunestrant
Number analyzed (Participants) | 45 | 20
Months | 11.07 [9.13 to NA] — Due to the high number of censored participants, there were not enough events to estimate the upper limit of the 95% confidence interval. | 10.02 [6.57 to 15.01]

11. Secondary Outcome: Percentage of Participants With Investigator-assessed Clinical Benefit Rate (CBR) (Between Arm C and Arm A)
Description: as for outcome 8
Time Frame: Randomization until measured progressive disease (up to 26 months)
Population: All participants who were randomly assigned to either arm A or arm C concurrently.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm C: Imlunestrant + Abemaciclib | Arm A: Imlunestrant
Number analyzed (Participants) | 213 | 213
Percentage of participants | 62.9 [56.4 to 69.4] | 44.1 [37.5 to 50.8]

12. Secondary Outcome: Time to Sustained Worsening of the "Worst Pain" as Measured by Worst Pain NRS (Between Arm A and Arm B)
Description: Time to sustained worsening of worst pain is defined as the time from randomization to the first increase (≥2 points) in the weekly average of the worst pain score, with confirmation in the next consecutive week. It was measured by the Worst Pain Numeric Rating Scale (NRS). NRS is a single-item, participant-administered, 11-point horizontal scale ranging from 0 to 10, with 0 representing "no pain" and 10 representing "pain as bad as you can imagine." Participants not known to have sustained worsening will be censored at the last documented assessment.
Time Frame: Randomization through follow-up (up to 24 months)
Population: All participants who were randomly assigned to either arm A or arm B and had at least one NRS assessment available (including censored). Number of participants censored in "Arm A=258," "Arm B=267."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 313 | 317
Months | NA [NA to NA] — Due to the high number of censored participants, there were not enough events to estimate the median and 95% confidence interval. | NA [NA to NA] — Due to the high number of censored participants, there were not enough events to estimate the median and 95% confidence interval.

13. Secondary Outcome: Time to Sustained Worsening of the "Worst Pain" as Measured by Worst Pain NRS (Between Arm C and Arm A)
Description: as for outcome 12
Time Frame: Randomization through follow-up (up to 20 months)
Population: All participants who were randomly assigned to either arm A or arm C concurrently and had at least one NRS assessment available (including censored). Number of participants censored in "Arm C=163," "Arm A=162."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Imlunestrant + Abemaciclib | Arm A: Imlunestrant
Number analyzed (Participants) | 204 | 198
Months | NA [NA to NA] — Due to the high number of censored participants, there were not enough events to estimate the median and 95% confidence interval. | NA [NA to NA] — Due to the high number of censored participants, there were not enough events to estimate the median and 95% confidence interval.

14. Secondary Outcome: Pharmacokinetics (PK): Plasma Concentration of Imlunestrant
Description: * Sampling timepoints for PK outcome analysis were relative to Imlunestrant dosing.
  * For Cycle 1 Day 1, sampling occurred at a "single" timepoint within the 2- to 4-hour window after Imlunestrant dosing, with the timepoint varying across analyzed participants.
Time Frame: Cycle 1 Day 1 (within 2 to 4 hours post-dose), Cycle 2 Day 1 (Predose), Cycle 3 Day 1 (3 hours post-dose, 5 hours post-dose), Cycle 4 Day 1 (Predose)
Population: All randomised participants who received at least 1 dose of study drug and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Arm A: Imlunestrant | Arm C: Imlunestrant + Abemaciclib
Number analyzed (Participants) | 276 | 189
nanograms per milliliter
  Cycle 1 Day 1 (within 2 to 4 hours postdose) | 45.7 (123) | 56.5 (122)
  Cycle 2 Day 1 (Predose): number analyzed (Participants) | 269 | 140
  Cycle 2 Day 1 (Predose) | 76 (76) | 64.9 (103)
  Cycle 3 Day 1 (3 hours post-dose): number analyzed (Participants) | 219 | 125
  Cycle 3 Day 1 (3 hours post-dose) | 141 (70) | 144 (73)
  Cycle 3 Day 1 (5 hours post-dose): number analyzed (Participants) | 209 | 123
  Cycle 3 Day 1 (5 hours post-dose) | 136 (69) | 146 (69)
  Cycle 4 Day 1 (Predose): number analyzed (Participants) | 178 | 105
  Cycle 4 Day 1 (Predose) | 85.2 (69) | 63 (97)

15. Secondary Outcome: Pharmacokinetics (PK): Plasma Concentration of Total Abemaciclib
Description: * Plasma concentration of total abemaciclib is the concentration of the parent abemaciclib and its metabolites in the plasma.
  * Sampling timepoints for PK outcome analysis were relative to Imlunestrant dosing.
  * For Cycle 1 Day 1, sampling occurred at a "single" timepoint within the 2- to 4-hour window after Imlunestrant dosing, with the timepoint varying across analyzed participants.
Time Frame: as for outcome 14
Population: All randomised participants who received at least 1 dose of study drug and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Arm C: Imlunestrant + Abemaciclib
Number analyzed (Participants) | 176
nanograms per milliliter
  Cycle 1 Day 1 (within 2 to 4 hours postdose) | 158 (120)
  Cycle 2 Day 1 (Predose): number analyzed (Participants) | 129
  Cycle 2 Day 1 (Predose) | 792 (82)
  Cycle 3 Day 1 (3 hours post-dose): number analyzed (Participants) | 100
  Cycle 3 Day 1 (3 hours post-dose) | 880 (74)
  Cycle 3 Day 1 (5 hours post-dose): number analyzed (Participants) | 100
  Cycle 3 Day 1 (5 hours post-dose) | 926 (64)
  Cycle 4 Day 1 (Predose): number analyzed (Participants) | 79
  Cycle 4 Day 1 (Predose) | 783 (59)

16. Secondary Outcome: Overall Survival (OS) in the ITT Population
Description: OS in the ITT population
Time Frame: Randomization until death from any cause (estimated as up to 5 years)
Reporting Status: Not Posted, anticipated posting 2028-05

17. Secondary Outcome: OS in the ESR1-mutation Detected Population
Description: OS in the ESR1-mutation detected population
Time Frame: Randomization until death from any cause (estimated as up to 5 years)
Reporting Status: Not Posted, anticipated posting 2028-05

18. Secondary Outcome: Blinded Independent Review Committee (BIRC) Assessed PFS in the ESR1-Mutation Detected Population (Between Arm A and Arm B)
Description: as for outcome 1
Time Frame: Randomization to the date of first documented progression of disease or death from any cause (up to 28 months)
Population: All participants who were randomly assigned to either arm A or arm B and had ESR1 mutations detected at baseline (including censored). Number of participants censored in "Arm A=64," "Arm B=47."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 138 | 118
Months | 7.43 [4.83 to 11.07] | 5.49 [3.84 to 6.70]

19. Secondary Outcome: Percentage of Participants With Investigator-assessed Objective Response Rate (ORR) in the ESR1-Mutation Detected Population (Between Arm A and Arm B)
Description: as for outcome 6
Time Frame: Randomization until measured progressive disease (up to 28 months)
Population: All participants who were randomly assigned to either arm A or arm B and had ESR1 mutations detected at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 138 | 118
Percentage of participants | 11.6 [6.3 to 16.9] | 5.9 [1.7 to 10.2]

20. Secondary Outcome: Investigator-assessed Duration of Response (DoR) in the ESR1-Mutation Detected Population (Between Arm A and Arm B)
Description: as for outcome 7
Time Frame: From Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up To 24 Months)
Population: All participants who were randomly assigned to either arm A or arm B, had ESR1 mutations detected at baseline and had achieved CR or PR responses (including censored). Number of participants censored in "Arm A=5," "Arm B=0."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 16 | 7
Months | 10.02 [3.98 to 14.59] | 5.59 [2.92 to 7.79]

21. Secondary Outcome: Percentage of Participants With Investigator-assessed Clinical Benefit Rate (CBR) in the ESR1-Mutation Detected Population (Between Arm A and Arm B)
Description: as for outcome 8
Time Frame: Randomization until measured progressive disease (up to 28 months)
Population: All participants who were randomly assigned to either arm A or arm B and had ESR1 mutations detected at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy
Number analyzed (Participants) | 138 | 118
Percentage of participants | 46.4 [38.1 to 54.7] | 36.4 [27.8 to 45.1]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 months
Description: Adverse events were reported for the "Safety Analysis Population."
Groups:
- Arm B: Investigator's Choice of Endocrine Therapy - Exemestane: This group includes Arm B participants for whom the Investigator's Choice of Endocrine Therapy was Exemestane. Participants received exemestane 25 mg administered orally once daily on days 1 to 28 of a 28-day cycle until disease progression or a criterion for discontinuation was met.
- Arm B: Investigator's Choice of Endocrine Therapy - Fulvestrant: This group includes Arm B participants for whom the Investigator's Choice of Endocrine Therapy was Fulvestrant. Participants received Fulvestrant 500 mg intramuscularly on days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond, until disease progression or a criterion for discontinuation was met.
Arm/Group | Arm A: Imlunestrant | Arm B: Investigator's Choice of Endocrine Therapy - Exemestane | Arm B: Investigator's Choice of Endocrine Therapy - Fulvestrant | Arm C: Imlunestrant + Abemaciclib
All-Cause Mortality (participants affected / at risk) | 62/327 | 8/32 | 82/292 | 36/208
Serious Adverse Events (participants affected / at risk) | 46/327 | 6/32 | 49/292 | 42/208
Other Adverse Events (participants affected / at risk) | 250/327 | 26/32 | 229/292 | 203/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Imlunestrant (N=327) | Arm B: Investigator's Choice of Endocrine Therapy - Exemestane (N=32) | Arm B: Investigator's Choice of Endocrine Therapy - Fulvestrant (N=292) | Arm C: Imlunestrant + Abemaciclib (N=208)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival papillae (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 3 (3) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 4 (4)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic reaction (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound treatment (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Imlunestrant (N=327) | Arm B: Investigator's Choice of Endocrine Therapy - Exemestane (N=32) | Arm B: Investigator's Choice of Endocrine Therapy - Fulvestrant (N=292) | Arm C: Imlunestrant + Abemaciclib (N=208)
Anaemia (Blood and lymphatic system disorders) | 38 (52) | 8 (11) | 45 (62) | 91 (128)
Leukopenia (Blood and lymphatic system disorders) | 7 (11) | 0 (0) | 7 (13) | 22 (32)
Neutropenia (Blood and lymphatic system disorders) | 10 (13) | 0 (0) | 5 (5) | 55 (111)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (8) | 0 (0) | 8 (8) | 20 (23)
Abdominal pain (Gastrointestinal disorders) | 20 (21) | 0 (0) | 10 (12) | 26 (32)
Abdominal pain upper (Gastrointestinal disorders) | 12 (14) | 1 (1) | 5 (5) | 17 (21)
Constipation (Gastrointestinal disorders) | 35 (38) | 3 (3) | 19 (22) | 15 (16)
Diarrhoea (Gastrointestinal disorders) | 71 (101) | 3 (3) | 37 (41) | 180 (372)
Nausea (Gastrointestinal disorders) | 59 (74) | 4 (4) | 39 (45) | 104 (144)
Vomiting (Gastrointestinal disorders) | 31 (44) | 1 (1) | 15 (17) | 66 (112)
Asthenia (General disorders) | 33 (39) | 5 (5) | 21 (23) | 35 (46)
Fatigue (General disorders) | 45 (48) | 2 (2) | 19 (19) | 46 (59)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 19 (21) | 0 (0)
Oedema peripheral (General disorders) | 11 (15) | 1 (1) | 8 (10) | 13 (13)
Pyrexia (General disorders) | 16 (20) | 1 (1) | 10 (10) | 14 (20)
Covid-19 (Infections and infestations) | 22 (24) | 2 (2) | 22 (23) | 11 (11)
Nasopharyngitis (Infections and infestations) | 7 (10) | 2 (2) | 9 (10) | 8 (8)
Urinary tract infection (Infections and infestations) | 11 (15) | 2 (2) | 21 (24) | 10 (12)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 41 (53) | 1 (1) | 43 (64) | 35 (49)
Aspartate aminotransferase increased (Investigations) | 47 (59) | 3 (3) | 46 (65) | 43 (55)
Blood alkaline phosphatase increased (Investigations) | 30 (41) | 1 (1) | 32 (47) | 14 (18)
Blood creatinine increased (Investigations) | 11 (20) | 1 (1) | 7 (10) | 44 (66)
Gamma-glutamyltransferase increased (Investigations) | 17 (23) | 1 (1) | 23 (28) | 5 (5)
Lymphocyte count decreased (Investigations) | 15 (27) | 0 (0) | 20 (34) | 9 (11)
Neutrophil count decreased (Investigations) | 10 (20) | 0 (0) | 15 (23) | 47 (89)
Platelet count decreased (Investigations) | 12 (22) | 0 (0) | 10 (17) | 18 (21)
Weight decreased (Investigations) | 12 (13) | 0 (0) | 15 (17) | 14 (16)
White blood cell count decreased (Investigations) | 14 (28) | 1 (1) | 17 (26) | 33 (67)
Decreased appetite (Metabolism and nutrition disorders) | 26 (31) | 1 (1) | 14 (15) | 42 (53)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (25) | 0 (0) | 21 (29) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 5 (7) | 19 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 (65) | 4 (5) | 43 (57) | 20 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 38 (47) | 1 (1) | 26 (30) | 12 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 3 (5) | 10 (11) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (19) | 3 (3) | 22 (24) | 9 (11)
Dizziness (Nervous system disorders) | 10 (11) | 1 (1) | 9 (9) | 12 (14)
Headache (Nervous system disorders) | 28 (30) | 2 (3) | 27 (28) | 20 (25)
Neuropathy peripheral (Nervous system disorders) | 7 (8) | 2 (2) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (35) | 2 (2) | 19 (21) | 18 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 1 (1) | 13 (15) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 5 (5) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 8 (10) | 10 (10)
Hot flush (Vascular disorders) | 22 (22) | 1 (1) | 20 (20) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT04975308/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT04975308/SAP_001.pdf